CLINICAL TRIAL: NCT01764802
Title: Psychosexual Intervention for Gynecologic and Breast Cancer Patients
Brief Title: Psychosexual Intervention in Patients With Stage I-III Gynecologic or Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kristen Carpenter, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-10077; NCI-2012-01341 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1R21CA149675-01A1 (NIH)
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Sarcoma; Ovarian Stromal Cancer; Stage I Uterine Sarcoma; Stage I Vaginal Cancer; Stage I Vulvar Cancer; Stage IA Cervical Cancer; Stage IA Endometrial Carcinoma; Stage IA Fallopian Tube Cancer; Stage IA Ovarian Epithelial Cancer; Stage IA Ovarian Germ Cell Tumor; Stage IA Primary Peritoneal Cavity Cancer; Stage IB Cervical Cancer; Stage IB Endometrial Carcinoma; Stage IB Fallopian Tube Cancer; Stage IB Ovarian Epithelial Cancer; Stage IB Ovarian Germ Cell Tumor; Stage IB Primary Peritoneal Cavity Cancer; Stage IC Fallopian Tube Cancer; Stage IC Ovarian Epithelial Cancer; Stage IC Ovarian Germ Cell Tumor; Stage IC Primary Peritoneal Cavity Cancer; Stage II Endometrial Carcinoma; Stage II Gestational Trophoblastic Tumor; Stage II Uterine Sarcoma; Stage II Vaginal Cancer; Stage II Vulvar Cancer; Stage IIA Cervical Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Epithelial Cancer; Stage IIA Ovarian Germ Cell Tumor; Stage IIA Primary Peritoneal Cavity Cancer; Stage IIB Cervical Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Epithelial Cancer; Stage IIB Ovarian Germ Cell Tumor; Stage IIB Primary Peritoneal Cavity Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Epithelial Cancer; Stage IIC Ovarian Germ Cell Tumor; Stage IIC Primary Peritoneal Cavity Cancer; Stage III Gestational Trophoblastic Tumor; Stage III Uterine Sarcoma; Stage III Vaginal Cancer; Stage III Vulvar Cancer; Stage IIIA Cervical Cancer; Stage IIIA Endometrial Carcinoma; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIA Primary Peritoneal Cavity Cancer; Stage IIIB Cervical Cancer; Stage IIIB Endometrial Carcinoma; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIB Primary Peritoneal Cavity Cancer; Stage IIIC Endometrial Carcinoma; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IIIC Primary Peritoneal Cavity Cancer; Breast Cancer
Keywords: Psychosexual Intervention; Cancer; Gynecologic Cancer; Breast Cancer
MeSH Terms: conditions — Vaginal Neoplasms; Vulvar Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Gestational Trophoblastic Disease; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (enhanced standard care) (Active Comparator): Patients participate in enhanced standard care intervention comprising stress reduction, information delivery regarding cancer treatments and sexuality delivered over two sessions.
  Interventions: Other: behavioral, psychological or informational intervention
- Arm II (psychological intervention) (Experimental): Patients participate in individual or group therapy over 1.5 hours weekly for 6 weeks, bi-weekly for 8 weeks, and monthly for 2 months and complete assessment interviews.
  Interventions: Other: behavioral, psychological or informational intervention

INTERVENTIONS:
Other: behavioral, psychological or informational intervention — Participate in enhanced standard care
  Arms: Arm I (enhanced standard care)
Other: behavioral, psychological or informational intervention — Participate in psychological intervention
  Arms: Arm II (psychological intervention)

SUMMARY:
This randomized phase II trial studies how well psychosexual intervention works in patients with stage I-III gynecologic or breast cancer. Psychosexual intervention may improve sexual and psychosocial function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Efficacy for reducing the severity of sexual distress, difficulty, and dysfunction in a phase II randomized clinical trial (RCT).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (Enhanced standard care): Patients participate in enhanced standard care intervention comprising stress reduction, information delivery regarding gynecologic or breast cancer treatments and sexuality, and provision of a survivorship care plan (SCP) created using OncoLink over 1 hour following baseline assessment and before 6 months.

ARM II (Psychological intervention): Patients participate in individual or group therapy over 1.5 hours weekly for 4 weeks, bi-weekly for 8 weeks, and monthly for 2 months and complete assessment interviews.

After completion of study treatment, patients are followed up at 3, 6, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III gynecologic (any site) or breast cancer
* Able to speak/read English
* Able to give informed consent

Exclusion Criteria:

* Prior non-gynecologic/breast cancer diagnosis
* Refusal of any cancer treatment(s)
* Non-ambulatory
* Concurrent diagnosis of organic brain syndrome, dementia, mental retardation, or significant sensory deficit
* Major mental illness (e.g, schizophrenia, major depressive disorder)
* Current/recent (prior 12 months) pregnancy
* Residence > 70 miles from research site

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Sexual behavior/repertoire (kissing, intercourse, etc.) graded using the Sexual Experiences Scale (SES) | Up to 2 months
  Multilevel modeling will be used to model time effects compared to repeated-measures analysis of variance (ANOVA) because it allows not only fitting different patterns of average change (i.e., linear, quadratic), but also estimates individual variability in the rate of change. Both linear and quadratic change models will be tested and an optimal model will be determined. 95% confidence intervals will be obtained.
Sexual responsiveness (desire, arousal, orgasm) using the Female Sexual Functioning Index (FSFI) | Up to 4 weeks
  Principal components analysis yields six subscales: desire, arousal, lubrication, orgasm, satisfaction, and pain. Items are rated using the Likert scales. 95% confidence intervals will be obtained.
Sexual satisfaction graded using the global evaluation from the Derogatis Sexual Function Inventory (DSFI) | Up to 2 months
  95% confidence intervals will be obtained.
Sexual distress graded using the female Sexual Distress Scale (FSDS) | Up to 4 weeks
  The Likert scale will be used. 95% confidence intervals will be obtained.
Sexual pain graded using the International Pelvic Pain Society Pelvic Pain Assessment, patient/physician version | Up to 9 months

SECONDARY OUTCOMES:
Emotional distress graded using the Profile of Mood States (POMS) | Up to 9 months
  The Likert scale will be used. 95% confidence intervals will be obtained.
Depressive symptoms graded using the Center for Epidemiologic Studies Depression Scale (CES-D) | Up to 9 months
  The Likert scale will be used. 95% confidence intervals will be obtained.
Health-related quality of life graded according to the RAND Medical Outcomes Study, Short-form 12 (SF-12) | Up to 9 months
  The eight primary subscales are summarized into two component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
Cancer-related stress graded according to the Impact of Events Scale-Revised (IES-R) | Up to 9 months
Body change stress graded according to the Impact of Treatment Scale (ITS) | Up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M. Carpenter, Ph.D, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Black LL, Conroy K, Lustberg M, Salani R, Andersen BL, Carpenter KM. Association of sexual pain and psychological factors among gynecologic and breast cancer patients: application of components of the fear-avoidance model of chronic pain. J Behav Med. 2025 Jun;48(3):536-543. doi: 10.1007/s10865-025-00560-3. Epub 2025 Mar 13. PMID 40082377
- See also: Jamesline — http://cancer.osu.edu